CLINICAL TRIAL: NCT04678154
Title: Evaluation of a New Strategy for Protocolized Antibiotic Care for Severe Open Fractures: SEXTANT - A Multicenter Randomized Control Trial
Brief Title: Evaluation of a New Strategy for Protocolized Antibiotic Care for Severe Open Fractures: SEXTANT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-19-2-0062
Record Dates: First submitted 2020-12-11; First posted 2020-12-21 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Surgical Site Infection
Keywords: Surgical site infection risk prevention; Bacterial species type and antibacterial sensitivities
MeSH Terms: interventions — Standard of Care; Vancomycin; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Participants in the control group will receive standard of care treatment for their injury, to include all institution specific standard treatment (prophylactic and otherwise) for preventing and treating infection.
  Interventions: Drug: Standard of care
- Treatment (Experimental): The patients in the SEXTANT cohort will have 1000 mg of Vancomycin and 1200 mg of Tobramycin administered to the wound surface, fracture site and exposed hardware (if any) just prior to suture closure of the wound or flap. The SEXTANT cohort will then receive at least 72 hours of systemic antibiotic therapy targeted to the modern wound bioburden.
  Interventions: Drug: Vancomycin and Tobramycin

INTERVENTIONS:
Drug: Standard of care — Participants in the control group will receive standard of care treatment for their injury, to include all institution specific standard treatment (prophylactic and otherwise) for preventing and treating infection.
  Arms: Control
Drug: Vancomycin and Tobramycin — The patients in the SEXTANT cohort will have 1000 mg of Vancomycin and 1200 mg of Tobramycin administered to the wound surface, fracture site and exposed hardware (if any) just prior to suture closure of the wound or flap. The SEXTANT cohort will then receive at least 72 hours of systemic antibiotic therapy targeted to the modern wound bioburden.
  Arms: Treatment

SUMMARY:
The proposed study is a multi-center, prospective randomized controlled trial comparing current standard of care treatment to the SEXTANT treatment protocol in patients with Type III open fractures of the tibia and IIIB fractures of the ankle and hindfoot.

DETAILED DESCRIPTION:
Specific Aim 1: To compare the surgical site infection (SSI) rates of the current severe open fracture antibiotic strategy to a revised SEXTANT treatment strategy designed to address the modern wound bioburden at the time of wound closure or coverage.

Specific Aim 2: To compare the terminal bioburden of the wounds at the time of definitive closure or coverage as sampled by standard tissue microbiology.

Specific Aim 3: To compare rates of antibiotic-related serious adverse events (SAEs) of the two treatment groups.

Exploratory Aim 4: To pilot the use of available and emerging rapid PCR platforms for wound pathogen identification in a sub-cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Injury meeting at least one of the following criteria:

   * Gustilo type III tibia (OTA 41 plateau, OTA 42 shaft and OTA 43 pilon) requiring a second procedure for final debridement and definitive coverage / closure following the index stabilization
   * Gustilo type IIIB ankle fractures (OTA 44)
   * Gustilo type IIIB calcaneus fractures (OTA 82)
   * Gustilo type IIIB talus fractures (OTA 81)
   * Traumatic "zone-of-injury" trans-tibial amputations requiring DPC, and/or flap coverage
2. Ages 18 - 64 years inclusive
3. Patients may have risk factors for infection including diabetes, immunosuppression from steroids or other medications, HIV, or other infections.
4. Patients may have a traumatic brain injury.
5. Patients may have other fractures including spine, upper extremity fractures, contralateral lower extremity injuries, ipsilateral pelvis, hip, femur or foot injuries.
6. Patients may be treated initially at an outside institution prior to transfer to the study institution, as long as the definitive wound closure or coverage was not performed prior to entrance into the study.
7. Patients with bilateral injuries that meet inclusion criteria may be included, but only the limb rated as "more severe" by the treating surgeon will be enrolled in the study.
8. Patients may have co-existing non-tibial or hindfoot infection, with or without antibiotic treatment.
9. Patients may be definitively stabilized using any method (nail, plate, ex fix or cast).
10. Patients may have a fasciotomy.

Exclusion Criteria:

1. Patient in current therapy for a wound, implant or fracture site infection related to the study site.
2. Patient likely to have difficulty maintaining follow-up, including:

   * Diagnosis of a severe psychiatric condition
   * Intellectually challenged without adequate family support
   * Resides outside of the hospital's catchment area
   * Planning to follow-up at another medical center
   * Being a prisoner
   * Not having a means of contact (address, cell phone, home phone, e-mail)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Deep surgical site infection | 182 days from injury
  To compare the surgical site infection (SSI) rates of the current severe open fracture antibiotic strategy to a revised SEXTANT treatment strategy designed to address the modern wound bioburden at the time of wound closure or coverage.

SECONDARY OUTCOMES:
Deep surgical site infection | 365 days from injury
  To compare the surgical site infection (SSI) rates of the current severe open fracture antibiotic strategy to a revised SEXTANT treatment strategy designed to address the modern wound bioburden at the time of wound closure or coverage.
Fracture revision rates | 365 days from injury
  Fracture revision rates for non-union, flap failure, amputation, the development of resistant bacteria discovered at revision surgery and antibiotic-related complications (C. difficile, nephrotoxicity, ototoxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Micahel J Bosse, MD, Principal Investigator — Carolinas Medical Center; Rachel Seymour, PhD, Principal Investigator — Atrium Health Musculoskeletal Institute Research; Renan C Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Anthony R Carlini, MS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (31):
- United States (31):
  - Stanford University, Redwood City, California
  - _University of California, San Francisco, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - St Mary's University/Tenent Health, West Palm Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Indiana University School of Medicine - Methodist Hospital, Indianapolis, Indiana
  - Indiana University/Eskenazi Health, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - LSU Health Sciences, New Orleans, Louisiana
  - University of Maryland , MD Department of Orthopaedics, Baltimore, Maryland
  - Walter Reed Military Medical Center, Bethesda, Maryland
  - Harvard/Mass General/Brigham Hospitals, Boston, Massachusetts
  - Hennepin County Medical Center / Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Jamaica Hospital Medical Center, Jamaica, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - METROHealth, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Temple University, Philadelphia, Pennsylvania
  - Brown University/Rhode Island Hospital, Providence, Rhode Island
  - Rhode Island Hospital/Brown University, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center - Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax MEdical Campus, Falls Church, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No